CLINICAL TRIAL: NCT01303289
Title: Clinical Evaluation of a Normoproteic Diet With Ultra High Temperature Treatment
Brief Title: Clinical Evaluation of a Normoproteic Diet
Acronym: STDUGR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vegenat, S.A. (Industry)
Responsible Party: África Jiménez Jiménez, VEGENAT, S.A.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: VEGENAT-TDP STD UGR; TDP STANDARD 2006 (Other: VEGENAT, S.A.)
Record Dates: First submitted 2011-02-17; First posted 2011-02-24 (Estimated); Last update posted 2011-02-24 (Estimated); Status verified 2011-02

CONDITIONS: Severe Insufficient Nutrition
Keywords: Total Enteral Nutrition; Severe insufficient nutrition; T-Diet plus Standard; Lipidic profile; Quality of life
MeSH Terms: interventions — Phentermine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): The group 1 will receive the experimental product T-Diet plus Standard for 3 months.
  Interventions: Dietary Supplement: T-Diet plus Standard
- Group 2 (Active Comparator): The group 2 will receive the control product Jevity (Abbott Laboratories) for 3 months.
  Interventions: Dietary Supplement: Jevity

INTERVENTIONS:
Dietary Supplement: T-Diet plus Standard — T-Diet plus Standard is a complete balanced protein and energy oral nutrition supplement, indicated for the dietary management of patients with related malnutrition.
  Other Names: TDP STD
  Arms: Group 1
Dietary Supplement: Jevity — JEVITY is a diet for tube-fed patients in the medium to long term, to varying degrees of malnutrition with gastrointestinal disorders.
  Other Names: JEV ABBT
  Arms: Group 2

SUMMARY:
The main objective of this trial is the clinical evaluation of a normoproteic diet, when this diet is used for total enteral nutrition in geriatric people.

For 3 months,all the participants in the study will receive only tube feeding: The experimental group will receive the commercial preparation to evaluate (T-Diet Plus ®, Vegenat SA) and the control group will receive a standard diet (Jevity ®, Abbott Laboratories).

DETAILED DESCRIPTION:
The project includes:

* Product tolerance study: gastrointestinal and metabolic complications related to the product administration.
* The monitoring of the intervention, and clinical and nutritional evaluation of the participants, including anthropometry, quality of life related to the health and clinical and nutritional status analytical evaluation (hematology and biochemistry).
* The determination of the major biochemical variables related to the lipid profile and assessment of the antioxidant defense system, and also certain markers of metabolic syndrome and associated cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 65 years old, of both sex, receiving total enteral nutrition by tube.
* Admitted to medically supervised institutions (homes, health centers).
* Requirement for total enteral nutrition standard, at least 3 months.
* Acceptance volunteer to participate in the study by signing the written informed consent (approved by the Ethics Committee of University Hospital Virgen de las Nieves).

Exclusion Criteria:

* Patients who receive drugs with lipid composition.
* Unstable clinical situation.
* Patients with terminal illness.
* Refusal or physical or mental inability to cooperate in the study.
* Participating in another study.
* Other causes: social causes, humanitarian, non-cooperation, etc..

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-02; Primary Completion 2007-01 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Nutritional status evaluation | 6 months
  Clinical evaluation of a comercial product: T-Diet Plus (normoproteic and specific diet), when is used for total enteral nutrition in geriatric people.

SECONDARY OUTCOMES:
Specific parameters measure | 6 months
  1. Confirm gastrointestinal and metabolic tolerance of the product.
  2. Consider the influence of the diet received on quality of life related to health.
  3. Study the changes in the nutritional status of elderly patients
  4. Assess changes in the lipid profile of patients
  5. Compare the evolution in blood levels of metabolic syndrome indicator parameters and other related to cardiovascular morbidity.
  6. Assess changes in the antioxidant defense system.

CONTACTS AND LOCATIONS:
Overall Officials: Ángel Gil, PhD, Principal Investigator — Departament of Biochemistry and Molecular Biology II. University of Granada
Locations (1):
- Department of Biochemistry and Molecular Biology II. University of Granada, Granada, Granada, Spain